CLINICAL TRIAL: NCT02017626
Title: FAST-Fish -Food Allergy Specific Treatment for Fish Allergy.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Professor, Dr. Med Hans-Joergen Malling, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K-489 DK
Record Dates: First submitted 2013-08-21; First posted 2013-12-23 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Fish Allergy
Keywords: Fish allergy; immunotherapy; hypoallergen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group 1 (Experimental): 5 patients will receive 10 single rising doses of mCyp c 1 (modified allergen)from 0.6 ng to 6 ug and two maintenance doses, and 2 patients will receive placebo
  Interventions: Biological: mCyp c 1
- Group 2 (Experimental): 6 patients will receive 10 single rising doses of mCyp c 1 from 6 ng to 60 ug and two maintenance doses, and two patients will receive placebo.
  Interventions: Biological: mCyp c 1

INTERVENTIONS:
Biological: mCyp c 1 — 2 patient groups with different doses of allergen.
  Other Names: A modified hypo-allergenic Parvalbumin

SUMMARY:
The aim of this study is to investigate the safety and tolerability of Subcutaneous Immunotherapy treatment (SCIT) with incremental doses of a modified recombinant fish parvalbumin (mCyp c 1) quantified in mass units:

To establish a safe dose of the candidate hypo-allergen in human subjects and To study the pharmaco-dynamics of the hypo-allergen administered to human subjects.

The study is performed as a placebo-controlled double-blinded randomized trial with 24 fish allergic patients allocated into three different groups of eight.

DETAILED DESCRIPTION:
The aim of the FAST project in general is to develop novel recombinant allergen-based therapeutics for the treatment of food allergy. The chosen approach is to modify recombinant allergens into hypo-allergenic molecules to decrease the risk of anaphylactic side-effects and to allow administration of higher doses leading to better efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject from 18 to 65 years old and in general good health as determined by past medical history and physical examination.
* Case history of allergy to fish ingestion.
* Specific IgE to fish by either a positive SPT to cod fish extract or an ImmunoCAP to cod fish above 0.70 kUA/L,(Class 2) at screening.
* Positive Double blind placebo-controlled Food challenge (DBPCFC) with fish within the last two years.
* FEV1 at least 80% of predicted values at screening.
* Subject accepting to comply fully with the protocol.
* For woman of child bearing potential:

  * a negative urine pregnancy test at screening visit,
  * subject must receive a medically effective contraceptive method during the study

Exclusion Criteria:

* Food Anaphylactic Reaction: anaphylactic shock due to fish intake.
* Specific IgE (ImmunoCAP) to fish parvalbumin (rCyp c 1) below 0.35 kUA/L
* Ongoing pollen Immunotherapy (SIT).
* Any clinical condition that contraindicates SIT (EAACI-guidelines).
* Any significant clinical condition that the investigators judged might hamper the patient's safety or the study outcomes, these diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease, immunological and endocrine disease.
* Ongoing treatment with betablockers or ACE-inhibitors.
* Impossibility for the patient to comply with the scheduled visits.
* Pregnancy or nursing.
* Uncontrolled asthma.
* Subject who have participated in a clinical trial within 3 months prior to this one.
* Subject with a history of drug or alcohol abuse.
* Investigators, co-investigators, as well as their children or spouses and all the study collaborators should not be enrolled in the study.
* Patients with concurrent allergy symptoms can be included if patients can manage without antihistamines during screening and treatments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety in the form of number and severity of adverse events | 1 year
  Safety is evaluated by number and severity of adverse events

SECONDARY OUTCOMES:
Specific IgE | 1 year
  To study the pharmaco-dynamics of the hypo-allergen administered to human subjects i.e. Specific IgE.
IgG4 | 1 year
  Immunologic parameter.
Skin Prick Test | 1 Year
  Pharmaco-dynamics of the hypo-allergen administered to human subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Joergen Malling, MD, Principal Investigator — Allergy Clinic, Gentofte University Hospital
Locations (1):
- Allergy Clinic, Gentofte Hospital, Hellerup, Denmark

REFERENCES:
- See also: FAST: Towards safe and effective subcutaneous immunotherapy of persistent life-threatening food allergies. — http://www.ncbi.nlm.nih.gov/pubmed/?term=FAST%3A+towards+safe+and+effective+subcutaneous+immunotherapy+of+persistent+food+allergies